CLINICAL TRIAL: NCT02788968
Title: Conflict Detection Development During the Reasoning
Acronym: DéCoR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Cyceron (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014-A00935-42
Record Dates: First submitted 2016-02-09; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
Keywords: Psychology and Cognitive Neuroscience of development; Adolescent and young adult healthy volunteers; Anatomical and functionally Magnetic Resonance Imaging (MRI); Conflict detection; Reasoning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adolescents (Other): MRI 11-15 years
  Interventions: Other: MRI
- Young adults (Experimental): MRI 19-25 years
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Conventional reasoning tasks in both " with" and "without" cognitive conflict and realized during an MRI

SUMMARY:
The study to explore the development of these abilities with age, and called "Development of the conflict detection during the reasoning - Decor" will take place at CYCERON center and will include two groups of 22 participants: adolescents and young adults (N = 44). More specifically, this study aims to compare the changes in the brain of adolescents and young adults when conducting reasoning tasks for which there may be a cognitive conflict. Both groups of participants then spend an MRI (Magnetic Resonance Imaging) focused on the brain and in which they will carry out two classic tasks covering the main areas of reasoning (probabilistic and economic). Each of these tasks will be manipulated to include, or not, of making information call intuition to create or not a conflict between the correct answer (logic, normative) and biased response (intuitive, heuristic). Because of the major implication of this brain region in cognitive inhibition processes [of intuitive answer], measured brain activity in the anterior cingulate cortex (ACC) during both tasks version "with" or "no" conflict will be compared between groups. To better understand the links between the development of the CCA from adolescence to adulthood and conflict detection, activity measurements will be correlated with a part in morphometric measurements taken from the same area (volume Substance Grise - SG; characteristics of cortical sulci) and secondly to cognitive measures (executive functions - inhibitory control). This cross-sectional study focused on two age groups: 11-15 years and 19-25 years. For each age group, the participation of men / boys and women / girls will be balanced up.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and educated adolescents aged 11-15 years
* boy or girl
* French mother tongue
* Handedness : right
* Having been informed by the teen booklet and given its written consent, and whose parents or legal guardian will be ( a) signed the informed consent sheet of the protocol
* Medical examinations , neurological, neuroradiological norma

or

* All healthy young adults aged 19-25 years at university level or in the workforce
* man or woman
* Level ≥ 12 years of study (bachelor level )
* Native language: French
* Handedness : right
* Signing of the informed consent of the protocol
* Medical examinations , neurological, neuroradiological norma

Exclusion Criteria:

* Does not meet the targeted age groups
* Presents against -indications to MRI (severe claustrophobia , foreign bodies cons -indicated )
* This chronic intake of alcohol or drugs
* Cognitive disorders who could testify sudden onset of a stroke ; a history of head injury with loss of consciousness for more than 1 hour , or encephalitis
* A neurological chronic condition , psychiatric, endocrine , hepatic and infectious
* Major disease history (diabetes, chronic lung disease, heart disorder, metabolic , hematologic , endocrine or immunological severe, cancer)
* A medication that may interfere with brain imaging measures ( psychotropics, hypnotics, anxiolytics , neuroleptics, anti -Parkinson , benzodiazepines, anti-inflammatory drugs , antiepileptics, antihistamines , analgesics and muscle relaxants central ) .
* Manual predominantly left (after the first phone call with the contact person of CYCERON ; see section 9.1)
* Color Blindness
* Inability to submit the study for geographical or psychiatric reasons
* Pregnant and lactating women

The following criteria are specific to the adolescent group :

* Has pervasive developmental disorders and / or acquisitions identified by parents or legal guardian and (or ) the teachers
* Parents or legal guardian are not affiliated to a system of social security
* Unaccompanied by parent (s) (s) or legal guardian during the visit to CYCERON center

The following criteria are specific to the group of young adults :

* Non- affiliated to a social security scheme
* Be protected adult

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
brain activity in the anterior cingulate cortex (ACC ) | Day 1
  measured brain activity in the anterior cingulate cortex (ACC ) of healthy volunteers aged 11 to 15 participants , and from 19 to 25 years over two classic version reasoning tasks "with" and "without" cognitive conflict and realized on an MRI

SECONDARY OUTCOMES:
the activity recorded in the whole brain | Day 1
  the activity recorded in the whole brain of healthy volunteers aged 11 to 15 participants , and 19 to 25 years in two classic version reasoning tasks "with" and "without" cognitive conflict and carried out during the examination MRI
response time | Day 1
  response time recorded version "with" versus "without" cognitive conflict , participants in healthy volunteers aged 11-15 and 19-25 years in two classic reasoning tasks performed during an MRI
brain activity measured in the CSF in two classic reasoning tasks | Day 1
  Compare brain activity measured in the CSF in two classic reasoning tasks in both " with" and "without" conflict for each of the healthy volunteers participating groups

CONTACTS AND LOCATIONS:
Overall Officials: Wym WN De Nyes, PhD, Study Director — Cyceron
Locations (1):
- CHU Caen, Caen, France